CLINICAL TRIAL: NCT03185117
Title: Opioid Consumption After Hospital Discharge in Orthopedic Surgery
Status: Terminated | Type: Observational
Why Stopped: Low patient retention rate
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Nicoleta Stoicea, Research Scientist/ Adj. Assistant Professor, Ohio State University
Other Study IDs: 2016H0219
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Opioid Use; Arthropathy of Knee; Arthropathy of Hip
Keywords: opioid consumption; postdischarge; major orthopedic surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: Adult patients scheduled to undergo a total knee arthroplasty or total hip arthroplasty, who give written informed consent to participate in the study.

SUMMARY:
At the Ohio State University, and across the country, surgical patients admitted to the hospital are over-prescribed a significant amount of opioid medications upon discharge to home. Recent studies reveal that a large percentage of patients prescribed opioid medications after surgery have approximately half of the prescribed medication left over. This study aims to evaluate reported opioid use after surgery in patients undergoing major orthopedic surgery in order to better approach the issue with current opioid use and abuse trends while still providing adequate medical care and pain management to patients

DETAILED DESCRIPTION:
After being discharged from the hospital, opioids are major source of pain relief for patients. Previous studies show that 71% of patients prescribed opioid medications after thoracic surgery admitted to taking half or less of their prescribed opioid medications. The analysis showed a correlation between the amount of opioids consumed during the patient hospitalization and after discharge. Goesling et al. surveyed patients with or without previous history of opioid use who underwent total knee arthroplasty (TKA) or total hip arthroplasty (THA). Both groups were followed for 6 months to document the "natural history" of opioid use postoperatively and post discharge. For patients with preoperative opioid use undergoing TKA, 88.5% were shown to be using opioids after 1 month, 48.2% after 3 months and 53.5% after 6 months. For patients considered opioid naïve undergoing TKA, 66.5% were shown to be using opioids after 1 month, 16.6% after 3 months and 8.2% after 6 months. For patients with preoperative opioid use undergoing THA, 63.9% were shown to be using opioids after 1 month, 37.8% after 3 months and 34.7% after 6 months. For patients considered opioid naïve undergoing THA, 22.5% were shown to be using opioids after 1 month, 4.4% after 3 months and 4.3% after 6 months.

This study is observational and involves consenting adult patients undergoing major orthopedic surgery to pre-operative assessments including the Self Administered Gerocognitive Exam (SAGE) questionnaire, a cognitive test to identify mild-moderate cognitive impairment, and collection of demographic data and medical history. Phone call follow-ups include assessments of post-discharge pain and opioid consumption, and completing verbally an adapted Activities of Daily Living questionnaire. No additional risks have been identified by participating in this study. Participants may not directly benefit from participating in this trial, but the data collected could provide valuable insight into the discrepancy between required opioid pain medications and opioid pain medication prescription for adequate pain management. This insight could then be applied to reevaluate post-discharge pain management procedures and standards of care, therefore curbing opioid use and abuse trends.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age and older, undergoing orthopedic procedures (hip or knee arthroplasty)
* Capable and willing to consent
* Participants literate in English language

Exclusion Criteria:

* History of drug and /or alcohol abuse/ dependency
* Ketamine use during hospitalization
* Illiteracy
* Presence of a clinically diagnosed major psychiatric condition such as bipolar disorder, uncontrolled major depression, schizophrenia
* Any condition that the principle investigator may disqualify the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients at the OSUMC, 18 years of age and older scheduled to undergo a total knee arthroplasty or total hip arthroplasty, who give written informed consent to participate in the study and who meet all inclusion and no exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
opioid consumption over time | once per week, up to six weeks after surgery
  The opioid medication (oral morphine equivalent) taken by the patients will be assessed every week until the sixth postoperative week, to compare it with the amount prescribed by the physicians

CONTACTS AND LOCATIONS:
Overall Officials: Nicoleta Stoicea, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Efforts will be made to keep patient information confidential. individual participant data will only be available to researchers who are approved by the Institutional Review Board (IRB) to participate in study enrollment, follow up and data analysis

REFERENCES:
- [Background] Bartels K, Mayes LM, Dingmann C, Bullard KJ, Hopfer CJ, Binswanger IA. Opioid Use and Storage Patterns by Patients after Hospital Discharge following Surgery. PLoS One. 2016 Jan 29;11(1):e0147972. doi: 10.1371/journal.pone.0147972. eCollection 2016. PMID 26824844
- [Background] Goesling J, Moser SE, Zaidi B, Hassett AL, Hilliard P, Hallstrom B, Clauw DJ, Brummett CM. Trends and predictors of opioid use after total knee and total hip arthroplasty. Pain. 2016 Jun;157(6):1259-1265. doi: 10.1097/j.pain.0000000000000516. PMID 26871536